CLINICAL TRIAL: NCT00091780
Title: Epidemiology of Breast Arterial Calcification
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1271; R21HL077123 (NIH)
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To test the hypothesis that breast arterial calcification (BAC) seen on mammograms can identify women with an increased risk of coronary artery disease (CAD).

DETAILED DESCRIPTION:
BACKGROUND:

The study hypothesis is that breast arterial calcification (BAC) seen on mammograms can identify women with an increased risk of coronary artery disease (CAD). Annual mammograms are now routinely obtained on nearly 70% of women over forty years of age. The nearly 40 million examinations performed every year could be used to evaluate for BAC without any additional cost or change in current mammographic techniques. Identification of women with BAC has potential to substantially decrease the rate of heart attack and sudden death due to CAD in asymptomatic women. Before BAC can be used in a clinical setting, the age-specific prevalence of BAC needs to be fully defined using state of the art mammographic techniques. BAC then needs to be compared with well understood CAD risk factors and measures of coronary atherosclerosis. While this could be accomplished in a prospective study, the same goals can be attained using data already acquired in the Epidemiology of Coronary Calcification (ECAC) Study.

The study uses existing data on 612 non-high risk, non-referred women who are participants in the community-based ECAC Study funded by NIH from 1991-2006. This database includes traditional and newer coronary artery disease (CAD) risk factors and the results of electron beam computed tomography (EBCT) examinations for CAC at a baseline examination. Most of the women also have had risk factors and CAC measured during a follow-up examination, on average, five years after baseline examinations. The women in the ECAC Study, who do not have a history of myocardial infarction (MI) or stroke, represent the full age range routinely evaluated with mammograms. Almost all these women have their usual care, including annual mammograms, in Rochester, Minnesota.

DESIGN NARRATIVE:

The ECAC study has been instrumental in establishing the distribution of presence and quantity of CAC as well as the predictors of CAC. The database includes clinical and laboratory assessments of CAD risk factors, results of EBCTs, and findings on physical examinations. It will ultimately include information on adverse clinical events. There are 612 female participants who had one or more mammograms during the 12-year history of that study. Many women had 10 or more mammograms. The study will evaluate all of these mammograms for BAC and compare the findings with information already in the database. The combination of newly acquired data from mammograms with the existing data allows this to be a very comprehensive study and still be completed in the two-year time period. The findings can then be used to help design a future study to prospectively evaluate the impact of instituting preventive and early therapeutic measures for CAD in asymptomatic women with the appropriate features of BAC on mammography.

ELIGIBILITY:
No eligibility criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Whaley — Mayo Clinic